CLINICAL TRIAL: NCT05204641
Title: Effect of Fecal Microbiota Transfer on Progression of Parkinson Disease
Acronym: EFFACE-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Human Biome Institute S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Fecal Microbiota Transplant
MeSH Terms: conditions — Parkinson Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota transplant (Active Comparator): Pretreatment with rifaximin 3x 400 mg PO for 5 days Fecal Microbiota Transfer from healthy donor during colonoscopy. Assessments in clinical scales: 30 days, 90 days, 180 days and 12 months: Unified Parkinson Disease Rating Scale, modified Constipation Assessment Scale, Parkinson Disease Questionnaire-39, Non- Motor Symptoms Questionnaire, Gastrointestinal Dysfunction Scale for Parkinson Disease.
  Assessment of levodopa/benserazide 200+50 mg tablet pharmacokinetics before and 30 days and 1 year after intervention
  Interventions: Biological: Fecal Microbiota Transfer provided by Human Biome Institute
- Autotransplant of patients microbiota (Placebo Comparator): Pretreatment with rifaximin 3x 400 mg PO for 5 days Administration of auto-FMT during colonoscopy Assessments in clinical scales: 30 days, 90 days, 180 days and 12 months: Unified Parkinson Disease Rating Scale, modified Constipation Assessment Scale, Parkinson Disease Questionnaire-39, Non- Motor Symptoms Questionnaire, Gastrointestinal Dysfunction Scale for Parkinson Disease. Assessment of levodopa/benserazide 200+50 mg tablet pharmacokinetics before and 30 days and 1 year after intervention
  Interventions: Biological: Fecal Microbiota Transfer provided by Human Biome Institute

INTERVENTIONS:
Biological: Fecal Microbiota Transfer provided by Human Biome Institute — Fecal Microbiota Transfer with colonoscopy
  Other Names: mBiotix; Fecal Microbiota Transplantation

SUMMARY:
The aim of the study is to assess impact of Fecal Microbiota Transfer (FMT) on clinical symptoms of Parkinson's disease. Assesment of tremor, slowness of movements and balance problems before and after FMT will be performed. The effect of FMT on frequency of constipations, which are common among Parkinson disease patients and have negative impact on quality of life and drug absorption will also be assessed. Detailed assessment of absorption of levodopa, which is the golden standard of treatment of Parkinson disease, is planned. It is planned to recruit 40 patients with diagnosis of Parkinson disease and indications for colonoscopy (constipations, age >50 years). Patients will be randomly assigned to the group receiving treatment with FMT or identically looking placebo. It will be administered to intestine during colonoscopy. Patients will be assessed by neurologist few times after the procedure. Psychological assessment and examination of gait and balance by physiotherapist is also planned. The last assessment will be performed after 12 months to see if the clinical effect can be observed for such a long time. The composition of the intestinal microbiota will be carefully assessed before and after the procedure in order to identify pathogens that may affect the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Consent to undergo colonoscopy

Exclusion Criteria:

* perforation or obstruction of gastroenteric tract,
* radiotherapy of abdomen or pelvis region
* severe heart, liver or kidney failure
* coagulation disorders
* immunity disorders
* current viral, bacterial or fungal infection
* abdominal aortic aneurysm qualifying for surgery, pregnancy and lactation treatment with Duodopa, deep brain stimulation or apomorphine
* colonoscopy confirmed colon polyps, except for lesions <5 mm qualified for the NBI International Colorectal Endoscopic I group or other potentially neoplastic lesions after evaluation in white light and narrow beam imaging (NBI)
* severe food allergy with a history of anaphylaxis after consumption of the product.
* microbiological stool evaluation with detection of: methicillin-resistant Staphylococcus aureus (MRSA), Klebsiella pneumoniae carbapenemase (KPC), metallo-β-lactamase (MBL), extended-spectrum beta-lactamase (ESBL), vancomycin-resistant Enterococci (VRE), Salmonella, Shigella, Yersinia. If any other atypical pathogen are to be detected in general stool culture, it will be assessed on an individual basis.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Change in progression of motor symptoms of Parkinson Diseae | 12 months
  Reduction or no change in Unified Parkinson Disease Rating Scale part III (motor) in off state (min. 0, max 108 points)

SECONDARY OUTCOMES:
Change in bowel movements | 0,1,3,6,12 months
  Change of score in Gastrointestinal Dysfunction Scale for Parkinson Disease ( a minimum score of 1 and a maximum score of 108)
Change in bowel movements | 0,1,3,6,12 months
  Change of score in modified Constipation Assessment Scale (a minimum score of 0 and a maximum score of 16)
Change in MDS- Non Motor Scale and subscales | 0,1,3,6,12 months
  Rater-completed assessment that measures frequency and severity of 13 non-motor domains, over 52 items and covers a range of key non-motor symptoms both PD and treatment related
MoCA change | It is a 30-point assessment that takes about 10 minutes to complete
  Detection of dementia symptoms. It is a 30-point assessment that takes about 10 minutes to complete with a physician.

OTHER OUTCOMES:
Change of levodopa bioavailability | 1 months, 12 months
  Change in levodopa-carbidopa concentration in peripheral blood (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Faculty of health sciences, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No